CLINICAL TRIAL: NCT06659549
Title: A Phase 2, Double-masked, Randomized, Multicenter, Parallel Group, Placebo-controlled Study to Investigate the Efficacy and Safety of GAL-101, 2%, Ophthalmic Solution in Patients With Non-foveal Geographic Atrophy Secondary to Non-neovascular Age-related Macular Degeneration: eDREAM Study
Brief Title: A Phase 2 Efficacy and Safety Study of GAL-101, 2% Ophthalmic Solution in Non-foveal Geographic Atrophy Secondary to Non-neovascular AMD
Acronym: eDREAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Galimedix Therapeutics Inc (Industry)
Collaborators: Lexitas Pharma Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GAL-101-C0201
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Geographic Atrophy of the Macula
Keywords: AMD; Geographic Atrophy; Age Related Macular Degeneration; Amyloid-Beta; Eye-drops
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Reading Centers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GAL-101 ophthalmic solution (Experimental): Patient will apply daily 2 eye drops of GAL-101 at 5 minutes interval
  Interventions: Drug: GAL-101
- Placebo (Placebo Comparator): Patient will apply daily 2 eye drops ofPlacebo at 5 minutes interval
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GAL-101 — Patient will apply daily 2 eye drops of GAL-101 at 5 minutes interval
  Arms: GAL-101 ophthalmic solution
Drug: Placebo — Patient will apply daily 2 eye drops of Placebo at 5 minutes interval
  Arms: Placebo

SUMMARY:
Age-related macular degeneration (AMD) affects millions of elderly patients. When advanced, there is Geographic Atrophy (GA) in the retina. This means that there is an area with a loss of light-sensitive cells, called photoreceptors. That part of the retina can no longer see. Atrophy begins as a small spot in the retina distant from the fovea which is the part of the retina responsible for sharp central vision. The GA grows, and when it reaches the fovea, vision is severely diminished, and details cannot be seen anymore. The purpose of the eDREAM study is to understand if GAL-101 can slow the growth of GA and prevent it from reaching the fovea. GAL-101 is given as eyedrops. eDREAM patients will administer study eyedrops every day. Patients will be assigned by chance (randomly) to receive either eye-drops that contain the new medication, GAL-101, or eyedrops without the active drug (Placebo). Neither patients nor doctors will know which treatment was assigned to each patient until the end of the study.

DETAILED DESCRIPTION:
In this study, if both eyes qualify for the study, the eye with the better BCVA will be defined as the study eye. If both eyes qualify for the study and have identical BCVA, then the eye with higher baseline peripheral retinal degenerations (PRD) will be defined as the study eye. If baseline PRD is identical, then the right eye (OD) will be defined as the study eye. Only the study eye will be dosed with the Investigation Medicinal Product (IMP).

During visits, patients will administer 3 applications of 1 drop of GAL-101 or a matching Placebo that does not contain the active pharmaceutical ingredient (API) at 5-minute intervals (i.e., 1st application, wait 5 minutes, 2nd application, wait 5 minutes, 3rd application), under the supervision of trained and authorized study personnel. In between visits, patients will be instructed to administer 2 applications of 1 drop at 5-minute intervals once a day.

The study will be comprised of a 12- to 24-month treatment period determined individually according to patients' overall placement in global study randomization. All patients will participate at least 12 months of treatment. The visit schedule includes the following: Screening visits (Visit 1a and 1b) for image capture and confirmation of study eligibility by a reading center; Baseline/Randomization/Day 1 (Visit 2); a phone call at 2 weeks; and on-treatment clinic visits for safety and efficacy evaluations at 1 month, 3 months, 6 months, 9 months, and 12 months. Patients will continue to attend on-treatment clinic visits at 3-month intervals after 12 months until the last patient randomized in the study has completed 12 months of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥55 years of age
* Willing and able to provide written informed consent
* Willing and able to comply with the study schedule and study assessments
* Able to successfully administer ophthalmic solution or have an appropriate designee (e.g., family member, health care professional) who can administer ophthalmic solution
* BCVA of ≥50 letters in the study eye using Early Treatment Diabetic Retinopathy Study (ETDRS) chart (i.e., 20/100 Snellen equivalent). Criterion will be confirmed at Baseline
* Refractive error between +3 and -6 diopters spherical equivalent in the study eye
* Sufficiently clear ocular media and adequate pupillary dilation to permit quality fundus imaging of the study eye, in the opinion of the Investigator. Criterion will be confirmed at Baseline
* Diagnosed with non-foveal GA secondary to non-neovascular AMD in the study eye, as confirmed by the reading center

  1. Well-delineated cumulative GA area between 1.25 and 12.0 mm2
  2. If GA is multifocal, at least 1 lesion ≥1.25 mm2
  3. GA lesions must be located outside a ≥100 µm radius from the center point of the fovea (i.e., this area must have intact retinal pigment epithelium [RPE] and outer retina)
  4. GA lesions must be located (partially or wholly) within a 2000 µm radius from the center point of the fovea
  5. GA lesions must be completely located within FAF imaging field (field 2 to 30-degree image centered on the fovea). GA lesion borders must be >300 µm from image edges
  6. GA lesions must be >300 µm from the optic disc and/or peripapillary atrophy
  7. Area of PRD must be cumulatively between 7.25 and 25.0 mm2

Exclusion Criteria:

1. Presence or history of choroidal neovascularization (CNV). Criterion will be confirmed at Baseline
2. History of laser therapy in the macular region, regardless of indication
3. History of herpes zoster
4. Ophthalmic disease or condition that requires or is likely to require surgery during the study period
5. GA with cumulative area <1.25 mm2
6. Any GA lesion within 100 µm radius from the center point of the fovea
7. Axial length >26 mm
8. Any ocular disease or condition other than non-neovascular AMD that may, in the opinion of the Investigator, interfere with study assessments, patient adherence to the study schedule, or interpretation of study data (e.g., epiretinal membrane, macular hole, glaucomatous optic neuropathy, etc.)
9. Intraocular surgery (including cataract extraction and crystalline lens replacement) within 3 months before Visit 1a or yttrium aluminum garnet (YAG) surgery within 2 months before Visit 1a, or planned either during the study period
10. Use of pegcetacoplan or avacincaptad pegol within 6 months before Visit 1a, or planned use during the study period
11. Use of any prescription or over-the-counter ophthalmic medication within 1 month before Visit 1a or planned use during the study period
12. Use of rigid contact lenses within 1 month before Visit 1a or planned use during the study period

    Non-study Eye:
13. BCVA of <5 letters using ETDRS chart (i.e., 20/800 Snellen equivalent)

    Either Eye:
14. History of uveitis
15. GA secondary to any condition other than non-neovascular AMD
16. History of active ocular infection or inflammation within 3 months before Visit 1a or Baseline. Criterion will be confirmed at Baseline
17. Underwent investigational treatment for AMD within 6 months before Visit 1a

    General Exclusion Criteria:
18. History of therapeutic radiation to the cranium
19. Known allergy or hypersensitivity to the investigational medicinal product (IMP) or any of its excipients
20. History of malignant disease
21. Use of hydroxychloroquine within 1 month before Visit 1a, or planned use during the study period
22. Participated or plan to participate in any other IMP study within 1 month before Visit 1a or during the study period
23. Use of lutein >10 mg per day or zeaxanthin >2 mg per day within 1 month before Visit 1a, or planned use during the study period
24. Any medical condition (including mental), in the opinion of the Investigator, that could interfere with study assessments, patient adherence to the study schedule, or interpretation of study data
25. Screening laboratory values, in the opinion of the Investigator, that make the patient unsuitable for study participation
26. Pregnant, nursing, or planning a pregnancy during the study. Criterion will be confirmed at Baseline
27. Unwilling or unable to use an acceptable method of contraception throughout the study if a woman of childbearing potential (WOCBP) or if a sexual partner of a WOCBP

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of GAL-101 ophthalmic solution in reducing the rate of change in GA lesion size. | From baseline to last on-treatment visit (48 up to 96 weeks)
  Comparison between groups of annual rate of change in the area of GA as measured by fundus autofluorescence (FAF).

SECONDARY OUTCOMES:
Efficacy of GAL-101 ophthalmic solution in reducing the rate of change in photoreceptor degeneration (PRD) in eyes with GA | From baseline to last on-treatment visit (48 up to 96 weeks)
  Comparison between groups of annual rate of change in the area of PRD as measured by optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (3):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
- Ophthalmological Center After S.V. Malayan, Yerevan, Armenia
- Centre Monticelli Paradis d'Ophtalmologie, Marseille, France
- Georgia (3):
  - Akhali Mzera Limited, Tbilisi
  - Caucasus Medical Centre LLC, Tbilisi
  - Chichua Medical Centre Mzera LLC, Tbilisi
- Universitäts-Augenklinik Bonn, Bonn, Germany
- Institute of Eye Surgery (IOES Waterford), Waterford, Ireland
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Medical Center, Tel Aviv
- Italy (2):
  - Medical Retina & Imaging Unit, IRCCS MultiMedica, Ospedale San Giuseppe, Milan, Milano
  - Unità di Oculistica, IRCCS Ospedale San Raffaele, Milan, Milano

IPD SHARING:
Plan to Share IPD: Undecided